CLINICAL TRIAL: NCT01443117
Title: Administration of Polysaccharide or Conjugated Pneumococcal Vaccines to HIV-Infected Pregnant Women: Safety and Magnitude, Persistence, and Transplacental Transfer of Vaccine-Serotype Pneumococcal Anti-Capsular Antibodies
Brief Title: Evaluating the Safety and Immune Response to Two Pneumococcal Vaccines in HIV-Infected Pregnant Women
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P1091; 11687 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pneumococcal Infections; HIV Infections
MeSH Terms: conditions — Pneumococcal Infections; HIV Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Step 1: PPV-23 Vaccine (Arm 1a) (Experimental): Participants will receive one intramuscular (IM) injection of 0.5 mL of the PPV-23 vaccine at baseline.
  Interventions: Biological: PPV-23 Vaccine
- Step 1: PCV-13 Vaccine (Arm 1b) (Experimental): Participants will receive one IM injection of 0.5 mL of the PCV-13 vaccine at baseline.
  Interventions: Biological: PCV-13 Vaccine
- Step 1: Placebo Vaccine (Arm 1c) (Placebo Comparator): Participants will receive one IM injection of 0.5 mL of the placebo vaccine at baseline.
  Interventions: Biological: Placebo Vaccine
- Step 2: PPV-23 Vaccine (Arm 2a) (Experimental): Participants will receive one IM injection of 0.5 mL of the PPV-23 vaccine 6 months after delivery.
  Interventions: Biological: PPV-23 Vaccine
- Step 2: PCV-13 Vaccine (Arm 2b) (Experimental): Participants will receive one IM injection of 0.5 mL of the PCV-13 vaccine 6 months after delivery.
  Interventions: Biological: PCV-13 Vaccine

INTERVENTIONS:
Biological: PPV-23 Vaccine — Administered as a 0.5 mL IM dose
  Arms: Step 1: PPV-23 Vaccine (Arm 1a); Step 2: PPV-23 Vaccine (Arm 2a)
Biological: PCV-13 Vaccine — Administered as a 0.5 mL IM dose
  Arms: Step 1: PCV-13 Vaccine (Arm 1b); Step 2: PCV-13 Vaccine (Arm 2b)
Biological: Placebo Vaccine — Administered as a 0.5 mL IM dose
  Arms: Step 1: Placebo Vaccine (Arm 1c)

SUMMARY:
HIV-infected people and pregnant women are at risk of developing severe pneumococcal disease. The purpose of this study is to compare the safety and immune response to two pneumococcal vaccines in HIV-infected pregnant women.

DETAILED DESCRIPTION:
Pneumococcus is the most common bacterial opportunistic infection in HIV-infected children, and it is the leading cause of bacterial pneumonias in HIV-infected pregnant and non-pregnant adults. Pneumococcal polysaccharide vaccine (PPV-23) and pneumococcal conjugate vaccine (PCV-13) are two vaccines used for the prevention of pneumococcal (PNC) disease. The PPV-23 vaccine is recommended by the Centers for Disease Control and Prevention (CDC) for HIV-infected adults, including HIV-infected pregnant women. The PCV-13 vaccine is recommended by the CDC for use in children, including HIV-infected children. Studies have shown that PCV-13 and vaccines like PCV-13 are safe for use in healthy pregnant women, but they have not been studied in HIV-infected pregnant women. This study will compare the safety and immune response to the PCV-13 and PPV-23 vaccines in HIV-infected pregnant women.

This study will enroll HIV-infected pregnant women in their second or third trimester who are receiving antiretroviral therapy. The study will take place in two steps. In Step 1, participants will be randomly assigned to receive PPV-23 vaccine, PCV-13 vaccine, or placebo vaccine. At a baseline study visit, participants will undergo a physical examination, medical history and nutritional status review, fetal heart rate measurement, blood collection, an ultrasound, an adherence questionnaire, and a nose and throat swab procedure. They will then receive their assigned vaccine. Participants will not be told which vaccine they are receiving. Participants will remain in the clinic for 30 to 60 minutes after receiving the vaccine for monitoring. They will attend study visits 14 to 21 days after the vaccination visit, at Week 8, and at the time of labor and delivery. During these visits, they will undergo select baseline study procedures. After delivery, participants' babies will have a physical examination and blood collection. At 2 and 4 months after delivery, participants' babies will undergo select baseline study procedures. Participants' babies will receive the PCV vaccine according to the local standard of care.

Step 2 of the study will begin 6 months after delivery, at which time participants and their babies will attend a study visit for a physical examination, medical history and nutritional status review, an adherence questionnaire, and blood collection. Participants who received the PPV-23 vaccine or the PCV-13 vaccine in Step 1 will end their participation in the study after this visit. Participants who received placebo vaccine in Step 1 will be randomly assigned to receive the PPV-23 vaccine or PCV-13 vaccine at this study visit but will not be told which vaccine they are receiving. Participants will attend a study visit 14 to 21 days after receiving the vaccine, which will include select study procedures.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* Pregnant women 18 to 39 years old who provide written informed consent prior to initiation of study
* Pregnant women 13 to less than 18 years old with a parent or legal guardian able and willing to provide signed informed consent or who have attained the minimum age of consent, as defined by the local Institutional Review Board (IRB), and who provide written informed consent prior to initiation of study
* Gestational age (greater than or equal to 15 weeks [15 weeks 0 days] to less than 33 weeks [32 weeks 6 days]) documented by the approximate date of the last menstrual period and corroborated by physical exam. Ultrasound will be performed at sites where it is available to confirm or correct gestational dates prior to immunization.
* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points. The same method may be used at both time points. All samples tested must be whole blood, serum, or plasma. More information on this criterion can be found in the protocol.
* Receipt of highly active antiretroviral therapy (HAART) for greater than or equal to 4 weeks prior to study entry; see World Health Organization (WHO) advice: http://www.who.int/hiv/pub/mtct/advice/en/index.html
* Documented platelet count of greater than 50,000/mm^3 and an absolute neutrophil count (ANC) of greater than 500/mm^3 less than or equal to 28 days prior to study entry
* Able to understand and comply with planned study procedures
* Women who are willing and able to comply with the study visits

Exclusion Criteria for Step 1:

* Receipt of PCV at any time prior to study entry documented by medical history or record
* Receipt of PPV-23 at any time prior to enrollment documented by medical history or record
* Receipt of any live licensed vaccine less than or equal to 4 weeks or inactivated licensed vaccine less than or equal to 2 weeks prior to study entry
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) less than or equal to 4 weeks prior to vaccination in this study, or expects to receive another non-licensed agent before delivery unless study approval is obtained
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 100.0 degrees Fahrenheit less than or equal to 24 hours prior to study entry
* Women who have virologic failure and ineffective ARV therapy as indicated by an increase in plasma HIV RNA copies/ml greater than 3-fold between initiation of HAART and the most recent prenatal visit
* Women who do not agree to be compliant with antiretroviral therapy during pregnancy
* Women who plan to terminate their pregnancy
* Women who have a documented prior history of stillbirth, persistent hypertension, preeclampsia, preterm premature rupture of the membranes less than 32 weeks gestation, oligohydramnios, lupus, HELP syndrome, or obstetric cholestasis
* Any women, who in the opinion of the investigator has a serious cardiovascular or pulmonary function disease and in whom a systemic reaction would pose a significant risk
* Use of anti-cancer systemic chemotherapy or radiation therapy less than or equal to 48 weeks prior to study entry, or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection)
* Ongoing neoplastic disease (excluding non-melanoma skin cancer, human papilloma virus [HPV]-related cervical dysplasia, and cervical intraepithelial neoplasia [CIN] Grades 1, 2, or 3)
* Long-term use of glucocorticoids, including oral or parenteral prednisone greater than or equal to 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 12 weeks of study entry, or high-dose inhaled steroids (greater than 800 mcg/day of beclomethasone dipropionate or equivalent) less than or equal to 12 weeks before study entry (nasal and topical steroids are allowed)
* Women who received corticosteroids for preterm labor less than or equal to 2 weeks before study entry
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) less than or equal to 12 weeks prior to study entry in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery
* Receipt of IL2, interferon (IFN), granulocyte-macrophage colony-stimulating factor (GMCSF) or other immune mediators less than or equal to 12 weeks before study entry
* Malaria during current pregnancy or other chronic disease (other than HIV) known to decrease transplacental transfer of antibodies
* Uncontrolled major psychiatric disorder
* History of a severe adverse reaction to inactivated polysaccharide or conjugated vaccines
* Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the person unable to meet the requirements of the study
* Pregnancy complications (in the current pregnancy) such as pre-term labor, hypertension (systolic blood pressure greater than or equal to 140 mm Hg and/or diastolic blood pressure greater than or equal to 90 mm Hg), and pre-eclampsia or any other pregnancy-related complication, which in the opinion of the investigator, might jeopardize the results of the study

Inclusion Criteria for Step 2:

* 24 weeks postpartum
* Completion of Step 1 of the study

Exclusion Criteria for Step 2:

* Pregnancy
* Receipt of any live licensed vaccine less than or equal to 4 weeks prior to entry or receipt of inactivated licensed vaccine less than or equal to 2 weeks prior to entry
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) less than or equal to 4 weeks prior to vaccination, or expects to receive another non-licensed agent within 30 days after vaccination
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 100.0 degrees Fahrenheit within 24 hours except when, in the opinion of the physician, withholding the agent entails even greater risk
* Use of anti-cancer systemic chemotherapy or radiation therapy or has developed immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection)
* Ongoing neoplastic disease (excluding non-melanoma skin cancer, human papilloma virus [HPV]-related cervical dysplasia, and cervical intraepithelial neoplasia [CIN] grades 1, 2, or 3)
* Use of glucocorticoids, including oral or parenteral prednisone greater than or equal to 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 2 weeks of entry in step 2. In some cases, entry in step can be delayed to avoid this exclusion criterion.
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) within 12 weeks prior to entry in step 2 or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during the 30 days following vaccination
* Receipt of IL2, interferon (IFN), granulocyte-macrophage colony-stimulating factor (GMCSF), or other immune mediators less than or equal to 12 weeks before entry in step 2

Ages: 13 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
For women: Grade 3 or higher adverse events | Measured through approximately 60 weeks
For women: Grade 3 or higher adverse events judged to be at least possibly related to the study treatment | Measured through approximately 60 weeks
For women: A 2-fold increase in ELISA or 4-fold rise in opsonic activity (OPA)-measured antibody concentrations | Measured at 14 to 21 days after immunization
  IgG antibodies to pneumococcal (PNC) 19A, 6B, 18C, and 5 will be measured by enzyme-linked immunosorbent assay (ELISA) and the capacity to opsonize to 19A and 6B will also be measured by OPA. The primary endpoint is a response to 3 out of 4 serotypes. A greater than or equal to 4-fold increase in OPA- and/or a greater than or equal to 2-fold increase in ELISA-measured IgG antibodies against PNC 19A and 6B will define a response against these serotypes. Responses to PNC 18C and 5 will rely only on the ELISA results.
For infants: ELISA-measured IgG antibody levels greater than or equal to 0.35ug/mL or OPA-measured antibody titers greater than or equal to 1:8 | Measured at 8 weeks of age for infants
  Reaching this level of antibodies for 3 of the 4 PNC serotypes that will be tested defines success
For women: Pneumonia or invasive pneumococcal disease | Measured through approximately 60 weeks
For women: Grade 3 or higher pregnancy-specific systemic adverse events | Measured through approximately 60 weeks
For women: Significant changes in HIV viral load in pregnant participants | Measured through approximately 60 weeks
For infants: Congenital defects | Measured through approximately 36 weeks
For infants: Pneumonia or invasive pneumococcal disease | Measured through approximately 36 weeks
For infants: In-utero or perinatal HIV infection | Measured through approximately 36 weeks
For infants: Immune interference with infant response to PCV vaccine | Measured through approximately 36 weeks

SECONDARY OUTCOMES:
Infant maternal antibodies at 2 months of life | Measured at 2 months of age for infants
Maternal and infant vitamin D levels | Measured through approximately 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Study Chair — University of Colorado, Denver

REFERENCES:
- [Background] Scott JA, Brooks WA, Peiris JS, Holtzman D, Mulholland EK. Pneumonia research to reduce childhood mortality in the developing world. J Clin Invest. 2008 Apr;118(4):1291-300. doi: 10.1172/JCI33947. PMID 18382741
- [Background] Lopez-Palomo C, Martin-Zamorano M, Benitez E, Fernandez-Gutierrez C, Guerrero F, Rodriguez-Iglesias M, Giron-Gonzalez JA. Pneumonia in HIV-infected patients in the HAART era: incidence, risk, and impact of the pneumococcal vaccination. J Med Virol. 2004 Apr;72(4):517-24. doi: 10.1002/jmv.20045. PMID 14981752